CLINICAL TRIAL: NCT02805699
Title: Beijing Municipal Science and Technology Commission
Brief Title: A Clinical Evaluation of Baofeikang Granule in Combined Pulmonary Fibrosis and Emphysema Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Principal Investigator, Cui Hongsheng, Director of Department of Respiration of Beijing University of Chinese Medicine Third Affiliated Hospital, Beijing Municipal Science & Technology Commission
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Z161100000516055
Record Dates: First submitted 2016-06-06; First posted 2016-06-20 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Combined Pulmonary Fibrosis and Emphysema
Keywords: Clinical Efficacy; Baofeikang Granules; Combined Pulmonary Fibrosis and Emphysema
MeSH Terms: conditions — Emphysema | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baofeikang Granule (Experimental): On the basis of comprehensive treatment of spasmolysis antiasthmatic and anti-inflammatory, expectorant,cough,give BaoFeikang Granules(by Beijing KangRentang Pharmaceutical Co., Ltd.), 1 bag, twice each day.
  Interventions: Drug: Baofeikang Granule
- Placebo (Placebo Comparator): On the basis of comprehensive treatment of spasmolysis antiasthmatic and anti-inflammatory, expectorant,coughand give Chinese medicine placebo (by Beijing Kang Rentang Pharmaceutical Co., Ltd., requirements and Chinese medicine BaoFeikang Granules in appearance and taste similar),1bag，twice each day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baofeikang Granule — To observe the efficacy and safety of Baofeikang granules on Combined Pulmonary Fibrosis and Emphysema Treatment.Baofeikang Granules consist of（Codonopsis 30g, Cordyceps fungi powder 12g, ophiopogon root 10g, Schisandra 10g, angelica 15g, Bulbus Fritillariae thunbergii 10g, Sophora flavescens 10g,Forsythia suspensa 12g，Pinellia 10g, saponins thorn 10g, Radix Peucedani 10g）.1 bags,P.O（Oral）twice of each 3 months cycle.
  Other Names: Treatment Group
  Arms: Baofeikang Granule
Drug: Placebo — On the basis of comprehensive treatment of spasmolysis antiasthmatic and anti-inflammatory, expectorant, cough ， give Chinese medicine placebo,1 bags,P.O（Oral）twice of each 3 months cycle.
  Other Names: Control Group
  Arms: Placebo

SUMMARY:
The purpose of this study is to confirm the efficacy and safety of BaofeiKang Granule in the treatment of Combined Pulmonary Fibrosis and Emphysema patients.

DETAILED DESCRIPTION:
A randomized, double blinded, placebo controlled study is conducted to observe the efficacy and safety of BaoFeiKang Granule in the treatment of patients with Combined Pulmonary Fibrosis and Emphysema. The Traditional Chinese Medicine（TCM） syndrome intergal,lung function ,Chronic Obstructive Pulmonary Disease Assessment Test（CAT）score, acute exacerbation, arterial blood gas analysis, chest High Resolution Computerized Tomography （HRCT）and liver and kidney function are to be calculated and tested before and after the trial.

1. Randomization All the selected cases is divided into the experimental group and the control group randomly, and the section size is 6. STATISTICAL ANALYSIS SYSTEM（SAS）statistical software are randomly assigned table，and clinical researchers given the corresponding code number to the selected qualified patients.According to the code number,patients receive the corresponding code number box.The persons who generate and preserve of tables are not involved in clinical trials.
2. Drug coding According to the protocol,the experimental duration of treatment is 3 months.The patients accept the medication for each month.
3. Blind method In the course of the study, the researchers and the subjects were not aware of the grouping of the research objects.
4. Sample size According to the formula,n=(Uα+Uβ)2*2P(1-P)/(P1-P0),the required sample size of each group is calculated.P1 represents for the efficiency of treatment group, P0 for the control group, P= (P1+P0) /2 * 100%;α＝0.05，β＝0.10，Uα=1.65，Uβ=1.28.According to the previous research results and literature research,P1=70%,P0=40%.It is calculated n = 47,and considering shedding rate of 20%,n =56.So actual each group includes 60 patients.
5. Implementation and management (1) training of 4 clinical researchers to master case collection methods and evaluation methods to minimize selection bias; (2) all experimental drugs are used in the same batch of drugs. (3) to collect data of the combination of medication and the treatment to exclude the impact of the above interference; (4) inform patients to get a more comprehensive evaluation and follow-up treatment.Special problems can get all respiratory department doctor's consultation, so as to achieve patient cooperation and understanding.(5)List the cases of loss or withdrawal, and specify the details and reasons.

ELIGIBILITY:
Inclusion Criteria:

1. conform to Combined Pulmonary Fibrosis and Emphysema Treatment diagnostic criteria;
2. conform to Qi and yin deficiency, phlegm and blood stasis syndrome diagnosis standard;
3. Patients with non acute episode;
4. Age between 45-75 (including 45 and 75);
5. signed the informed consent.

Exclusion Criteria:

1. Combined upper and lower respiratory infection, pulmonary tuberculosis, lung cancer or other lung diseases;
2. Combined with diabetes, cardiovascular, liver, kidney or hematopoietic system diseases, psychiatric patients;
3. Pregnancy and lactation patients;
4. Allergic to the subjects of the medicine.

Rejection criteria:

1. do not meet the inclusion criteria after entering the group;
2. the discovery of serious physical illness after entering the group;
3. do not follow the program medication of patients;

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in the efficacy of TCM syndrome index at 3 months | Baseline and 3 months after the start of treatment
  Observe the changes of the symptoms of wheezing, chest congestion, cough, shortness of breath and etc

SECONDARY OUTCOMES:
Changes from baselines in Chronic Obstructive Pulmonary Disease Assessment Test(CAT)at 3 months | Baseline and 3 months after the start of treatment
Changes from baselines in Arterial blood gas analysis(ABG)at 3 months | Baseline and 3 months after the start of treatment
The scope and degree of fibrosis and emphysema of pulmonary in chest High Resolution Computerized Tomography(HRCT) | Baseline and 3 months after the start of treatment
Changes from baselines in frequence of acute exacerbation of cough,sputum,dyspnea at 1,2,3 months | Baseline and 1，2，3 months after the start of treatment
  acute exacerbation defined as involving symptoms lasting for >2 days , leading to treatment with systemic glucocorticoids, antibiotics, hospitalization or emergency
Forced Expiratory Volume in one second(FEV1) | Baseline and 3 months after the start of treatment
  pulmonary function
Forced Vital Capacity(FVC) | Baseline and 3 months after the start of treatment
  pulmonary function
Total Lung Capacity(TLC) | Baseline and 3 months after the start of treatment
  pulmonary function
Diffusion capacity for Carbon monoxide of the Lung(DLCO) | Baseline and 3 months after the start of treatment
  pulmonary function

OTHER OUTCOMES:
Number of participants with adverse events | Before treatment and 1，2，3 months after the start of treatment
  Blood routine examination,Liver and Renal function,Electrocardiogram
Chronic Obstructive Pulmonary Disease Assessment Test(CAT) | 1，3，6 months after the course of treatment
  This is the follow-up index.
frequence of acute exacerbation of cough,sputum,dyspnea | 1，3，6 months after the course of treatment
  This is the follow-up index.

CONTACTS AND LOCATIONS:
Overall Officials: hongsheng cui, Ph.D，Professor, Study Chair — The Third Affiliated Hospital of Beijing University of Chinese Medicine; weibo Bi, Master, Principal Investigator — The Third Affiliated Hospital of Beijing University of Chinese Medicine; jianjun Wu, Master, Principal Investigator — The Third Affiliated Hospital of Beijing University of Chinese Medicine; ruifeng Jin, Master, Principal Investigator — The Third Affiliated Hospital of Beijing University of Chinese Medicine; chang'an Li, Master, Principal Investigator — The Third Affiliated Hospital of Beijing University of Chinese Medicine; minmin Shan, Master, Principal Investigator — The Third Affiliated Hospital of Beijing University of Chinese Medicine; qiuyi Chen, Bachelor, Principal Investigator — The Third Affiliated Hospital of Beijing University of Chinese Medicine; shengtao li, Bachelor, Principal Investigator — The Third Affiliated Hospital of Beijing University of Chinese Medicine
Locations (2):
- China (2):
  - Beijing University of Chinese Medicine Third Affiliated Hospital, Beijing, Beijing Municipality
  - Dongzhimen hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Yes